CLINICAL TRIAL: NCT06267183
Title: A Phase I, Single-center, Randomized, Double-blind, Single-dose, Dose-ascending, Placebo-controlled Clinical Study to Evaluate Safety, Tolerability and Pharmacokinetics of SV001 in Chinese Healthy Adult Volunteers.
Brief Title: A Clinical Study to Evaluate Safety, Tolerability and Pharmacokinetics of SV001 in Chinese Healthy Adult Volunteers.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Synvida Biotechnology Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SV001-101
Record Dates: First submitted 2024-02-01; First posted 2024-02-20 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SV001 (Experimental)
  Interventions: Drug: SV001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SV001 — SV001 ： single-dose
  Arms: SV001
Drug: Placebo — Placebo ： single-dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, PK and immunogenicity of SV001 compare to placebo in Chinese healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must fully understand the purpose, characteristics, methods and possible adverse reactions of the trial, volunteer as a subject, and sign the Informed Consent Form;
2. Subjects must have a Body Mass Index in the range of 19~26 kg/m2, with males weighted not less than 50 kg, and females weighted not less than 45 kg;
3. Subjects must be in good health as judged by the investigator.
4. Reliable contraception must be assured during and for some time after the trial.

Exclusion Criteria:

1. Subjects with a history of drug or other substance anaphylaxis;
2. Subjects with respiratory symptoms or abnormal respiratory tract;
3. Subjects currently having an oral disease that the investigator judged may affect use of the trial drug and devices;
4. Subjects with other diseases or factors with abnormal clinical manifestations;
5. Subjects having a history of drug abuse in the past or having used narcotics in the period prior to screening, or having a positive result in urine narcotics test at baseline period;
6. Subjects who smoked more than 5 cigarettes a day in the period before screening;
7. Subjects who consumed more than 14 units of alcohol per week in the period prior to screening, or who is positive in breath alcohol test at baseline period;
8. Subjects who have suffered a clinically significant severe disease or undergone major surgical operations within a certain period of time prior to receiving the investigational drug, or who are expected to require major operations during the clinical trial;
9. Subjects who used other drugs within a certain period of time before receiving the investigational drug;
10. Screening period: FEV1≤80% predicted value or FVC≤80% predicted value;
11. Subjects who have antibody positive for Human Immunodeficiency Virus, Hepatitis B surface antigen, Hepatitis C or Treponema Pallidum.
12. Subjects who have difficulty in venous blood collection or have a history of acupuncture syncope and blood phobia;
13. Female subjects who are tested positive for pregnancy during the screening or baseline period or are in lactation period;
14. Subjects who have participated in other drug clinical trials and used other drugs in clinical trials within a certain period of time before receiving the investigational drug;
15. Subjects who have a history of blood donation or blood loss of more than 400 mL in the period prior to screening;
16. Any other status in which the investigator deems inappropriate to participate in the present study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Approximately 1 years
  Adverse event type, incidence, duration

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Approximately 1 years
  PK (Pharmacokinetics)
Peak time（Tmax） | Approximately 1 years
  PK (Pharmacokinetics)
Area under the plasma concentration versus time curve (AUC) | Approximately 1 years
  PK (Pharmacokinetics)
half-life（T1/2） | Approximately 1 years
  PK (Pharmacokinetics)
Immunogenicity | Approximately 1 years
  ADA（Anti-drug antibody）

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, China